CLINICAL TRIAL: NCT02230514
Title: A Phase IIa, Single Center, Prospective, Randomized, Parallel, Two-arms, Single-dose, Open-label With Blinded Assessor Pilot Clinical Trial to Assess ex Vivo Expanded Adult Autologous Mesenchymal Stromal Cells Fixed in Allogeneic Bone Tissue (XCEL-MT-OSTEO-ALPHA) in Non Hypertrophic Pseudoarthrosis of Long Bones
Brief Title: Mesenchymal Stromal Cells for the Treatment of Non-union Fractures of Long Bones
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Hospital ASEPEYO Sant Cugat (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XCEL-PSART-01; 2013-005025-23 (EudraCT Number)
Record Dates: First submitted 2014-07-17; First posted 2014-09-03 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Atrophic Nonunion of Fracture
Keywords: Nonunion fracture; Long bones; Pseudoarthrosis; Cell therapy; Tissue engineering; Mesenchymal stromal cells
MeSH Terms: conditions — Fractures, Ununited; Pseudarthrosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Radiologist will assess images in a blinded manner
Oversight: Data Monitoring Committee: No

ARMS (2):
- XCEL-MT-OSTEO-ALPHA and surgery (Experimental): "ex-vivo" expanded autologous mesenchymal stromal cells fixed in allogenic bone tissue
  Interventions: Drug: XCEL-MT-OSTEO-ALPHA; Procedure: Surgery
- Autologous iliac crest and surgery (Other): Standard treatment
  Interventions: Other: autologous iliac crest; Procedure: Surgery

INTERVENTIONS:
Drug: XCEL-MT-OSTEO-ALPHA — "ex-vivo" expanded autologous mesenchymal stromal cells fixed in allogenic bone tissue in association with open surgery
  Arms: XCEL-MT-OSTEO-ALPHA and surgery
Other: autologous iliac crest — Autologous iliac crest in association with surgery
  Arms: Autologous iliac crest and surgery
Procedure: Surgery — Standard surgery for non-union fractures

SUMMARY:
The present study evaluates the effect of XCEL-MT-OSTEO-ALPHA in non-union fractures (pseudoarthrosis) of long bones in comparison to the standard treatment of autologous iliac crest.

XCEL-MT-OSTEO-ALPHA is a tissue engineering product composed by "ex-vivo" expanded autologous mesenchymal stromal cells fixed in allogenic bone tissue, produced by Xcelia (Blood and Tissue Bank of Catalonia).

The working hypothesis proposes that the tissue engineering is a valid and useful technique to achieve bone regeneration up to consolidation of non-union fractures.

DETAILED DESCRIPTION:
A phase IIa, single center, prospective, randomized, parallel, two-arms, single-dose, open-label with blinded assessor pilot clinical trial to assess ex vivo expanded adult autologous mesenchymal stromal cells fixed in allogeneic bone tissue (XCEL-MT-OSTEO-ALPHA) in non hypertrophic pseudoarthrosis of long bones.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years of age (male and female)
* Atrophic or hypotrophic metaphyseal-diaphyseal pseudarthrosis of long bones, confirmed radiographically.
* Signed Informed Consent Form
* The patient is able to understand the nature of the study

Exclusion Criteria:

* Suspicious of pseudarthrosis focus infection diagnosed by clinical inspection and blood analysis.
* Positive serology for HIV (Anti-HIV I/II-Ac), Hepatitis B (HBsAg, HBcAc), Hepatitis C (Anti-HCV-Ac) or Syphilis Lúes (TP-Ac).
* Significant abnormal laboratory tests that contraindicates patient's participation in the study.
* Pregnant woman or without proper anticonceptive measures according to the investigator, or breath feeding
* Smoker of more than 15 cigarettes a day
* Congenital disorders of bones (hypophosphatemia), bone metabolic disorders associated to primary or secondary hypoparathyroidism.
* Badly managed diabetes mellitus.
* Patients diagnosed with peripheral arterial disorders
* Previous therapeutic radiation (5 previous years) of the affected bone.
* Neoplasia within the previous 5 years, or without remission
* The patient is legally dependent
* Participation in another clinical trial or treated with an investigational medicinal product the previous 30 days
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria
* The patient does not accept to be followed-up for a period that could exceed the clinical trial length

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment of XCEL-MT-OSTEO-ALPHA in non-union fractures by imaging procedures | 12 month
  Hounsfield units quantification by tomography in both treatment arms

SECONDARY OUTCOMES:
Safety assessment of XCEL-MT-OSTEO-ALPHA in non-union fractures | 12 month
  Safety will be assessed by collecting adverse events throughout the experimental phase which includes a follow-up of 12 month.
Efficacy assessment of XCEL-MT-OSTEO-ALPHA in non-union fractures by imaging procedures | 6 month
  Characteristics of the callus by tomography and Characteristics of the callus by standard x-ray in both treatment arms
Efficacy assessment by quality of life test | 12 month
  Quality of life will be measured by EUROQOL-5D test

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Granell, MD, PhD, Principal Investigator — Hospital ASEPEYO Sant Cugat
Locations (1):
- Hospital ASEPEYO Sant Cugat, Sant Cugat del Vallès, Barcelona, Spain

REFERENCES:
- See also: Banc de Sang i Teixits (Blood and Tissue Bank of Catalonia) — http://www.bancsang.net/
- See also: Hospital ASEPEYO Sant Cugat — http://www.asepeyo.es/hospital-sant-cugat